CLINICAL TRIAL: NCT07130097
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE DOSE, CROSSOVER, PIVOTAL BIOEQUIVALENCE STUDY TO COMPARE ATIRMOCICLIB (PF-07220060) HIGHER DRUG LOAD IR MST TABLETS AND ATIRMOCICLIB IR MST TABLETS ADMINISTERED UNDER FED CONDITIONS IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Compare Two Tablet Formulations of Study Medicine Atirmociclib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4391009
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participant
Keywords: Healthy Participants, ,; Bioequivalence; Bioavailability; Pharmacokinetics; Tablet Formulation; Crossover Study; ADME (Absorption, Distribution, Metabolism, Elimination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A; Treatment Sequence A (Experimental): Single Oral Dose of reference tablet formulation PF-07220060, then at least 7 day washout, followed by a single oral dose of test tablet formulation PF-07220060
  Interventions: Drug: PF-07220060
- Regimen B; Treatment Sequence B (Experimental): Single Oral Dose of test tablet formulation PF-07220060, then at least 7 day washout, followed by a single oral dose of reference tablet formulation PF-07220060
  Interventions: Drug: PF-07220060

INTERVENTIONS:
Drug: PF-07220060 — Cyclin-dependent kinase-4 inhibitor
  Other Names: Atirmociclib

SUMMARY:
The purpose of this study is to understand bioequivalence (medicines that may have different names or be made in different ways, but have the same effect on the body) of the current PF-07220060 tablet formulation and the proposed higher drug load tablet that is already available in the market.

The study is seeking participants who are:

* Healthy males and females aged 18 to 65 years
* Willing and able to comply with all scheduled visits, treatment plan, lifestyle considerations, and other study procedures.
* Body Mass Index of 17.5-30.5 kilogram per meter squared (kg/m2); and a total body weight of more than 50 kilograms (kg) [110 pounds (lb)].

Participants in the study will receive a single dose of PF-07220060 by mouth after a meal, following at least 7 days, the participant will then receive another dose of PF-07220060. Each dose received by the participant will be a different tablet formulation, and the sequence of tablet formulations given will be random (just like a flipside of the coin).

The study will help the team understand how the difference in tablet formulation may, or may not, affect how the medicine is absorbed, processed, and removed by the body.

Participants will remain in the study clinic for at least 13 days and will have one follow-up contact.

ELIGIBILITY:
Inclusion:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.
* BMI of 17.5-30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Evidence of a personally signed and dated ICD indicating that the participant has been informed of all pertinent aspects of the study.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Exclusion:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* A positive urine drug test
* Unwilling or unable to comply with the Lifestyle Considerations criteria of this study
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2025-08-14 (Actual); Primary Completion 2025-10-26 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Area under the Plasma Concentration-Time profile from time 0 to time of last quantifiable data point (AUClast)) of test and reference atirmociclib formulations after a high fat/high calorie meal (If data does not permit AUCinf) | Pre-dose, 0, 0.5, 0.75, 1, 1.5, 2, 3, 4 ,6 , 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post dose in period 1 and period 2
  AUClast was area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (If data does not permit reporting of AUCinf). The geometric coefficient of variation is expressed in percentage. The ratio (Test/Reference) of adjusted means and 90% CI are then expressed as percentages.
Area under the Plasma Concentration-Time profile (AUC) from time 0 extrapolated to extrapolated infinite time (AUCinf) of test and reference atirmociclib formulations after a high fat/high calorie meal (If data permits). | Pre-dose, 0, 0.5, 0.75, 1, 1.5, 2, 3, 4 ,6 , 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post dose in period 1 and period 2
  AUCinf was area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf , if data permits). It is obtained from AUC (0-t) plus AUC (t-inf). The geometric coefficient of variation is expressed in percentage. The ratio (Test/Reference) of adjusted means and 90% CI are then expressed as percentages.
Maximum Observed Plasma Concentration (Cmax) profile of test and reference atirmociclib formulations after a high fat/high calorie meal | Pre-dose, 0, 0.5, 0.75, 1, 1.5, 2, 3, 4 ,6 , 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post dose in period 1 and period 2
  Cmax was the maximum observed plasma concentration directly observed from data. The geometric coefficient of variation is expressed in percentage. The ratio (Test/Reference) of adjusted means and 90% CI are then expressed as percentages.

SECONDARY OUTCOMES:
Number of Participants with Clinically Significant Abnormalities in Laboratory Parameters | From baseline up to 36 days after the last dose of study intervention (up to Day 36 post dose in period 2)
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | From baseline up to 36 days after the last dose of study intervention (up to Day 36 post dose in period 2)
Number of Participants with Clinically Significant Abnormalities in Vital Signs | From baseline up to 36 days after the last dose of study intervention (up to Day 36 post dose in period 2)
Number of Participants with Clinically Significant Electrocardiogram (ECG) Abnormalities | From baseline up to 36 days after the last dose of study intervention (up to Day 36 post dose in period 2)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4391009